CLINICAL TRIAL: NCT03559829
Title: Feasibility of Home-based Virtual Reality Rehabilitation for the Upper Extremity in Subacute and Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: NEOFECT Rehabilitation Solutions (Other)
Responsible Party: Principal Investigator, Maarten Lansberg, Associate Professor, Neurology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 37580; 125802 (Other: Stanford)
Record Dates: First submitted 2018-06-01; First posted 2018-06-18 (Actual); Results first posted 2019-05-01 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Arm - Intervention arm (Experimental): RAPAEL Smart Glove Arm The participant will be issued a Smart Glove and a tablet preloaded with the game software. The available games provide various kinds of motion tasks such as ADL-related tasks presented in an entertaining manner. The learning schedule algorithm automatically adjusts to the optimal level of difficulty to balance challenge and motivation. The participant will be expected to use the Smart Glove at home for 60 min per day for at least 5 days per week.
  Interventions: Device: RAPAEL Smart Glove

INTERVENTIONS:
Device: RAPAEL Smart Glove — The RAPAEL Smart Glove is a commercially available, non-invasive biofeedback based system for distal upper extremity rehabilitation. The Smart Glove is very lightweight and allows for easy movement of all distal upper extremity joints. It is made of an elastomer material that is simple to maintain and clean. The Bending Sensor is a variable resistor that changes as it is bent. The sensor is a 9-axis movement and position sensor that consists of 3 acceleration channels, 3 angular rate channels, and 3 magnetic field channels that measure wrist movements. They are connected to a computer system which can accurately compute the amount of individual finger movements.

SUMMARY:
Regaining upper extremity function is very important for stroke survivors to increase their independence and ability to perform activities of daily living (ADLs). Outpatient stroke rehabilitation currently takes place in a therapy clinic, however access can be limited by financial resources and transportation difficulties.

The Feasibility of Home-Based Virtual Reality Rehabilitation for the Upper Extremity in Subacute and Chronic Stroke Study seeks to explore the safety, usability, and efficacy of a home based virtual reality biofeedback system to promote distal upper extremity (wrist and hand) recovery after stroke. The purpose of the study is to assess the feasibility of using a home-based virtual reality system to increase the dose of upper extremity rehabilitation in subacute and chronic stroke patients.

DETAILED DESCRIPTION:
In this pilot study, we propose to test a virtual reality home-based intervention as an alternative or supplement to traditional rehabilitation for upper extremity weakness after stroke. We are hoping to discover that the device is easily adopted by patients and increases the dose of rehabilitation, as well as potentially leads to motor recovery.

With the increasing affordability and accessibility of virtual reality (VR) systems, VR has emerged as a new platform for stroke rehabilitation. VR therapy involves using computer-based programs to simulate daily tasks and events. VR has shown promise in both allowing patients to practice activities that directly translate to their ADLs, as well as motivating them by providing a novel and interesting virtual environment.

Relevance Regaining upper extremity function is very important for stroke survivors to increase their independence and ability to perform ADLs. The large majority of outpatient stroke rehabilitation currently takes place in a therapy clinic, however access is often limited by resource allocation, financial hardship, and transportation difficulties. The Smart Glove can provide an inexpensive and convenient means for stroke patients to continue their rehabilitation in the comfort of their own home.

Patient Population Subacute and chronic stroke patients presenting with upper extremity weakness, as identified by Stanford physicians in clinic, will be eligible for participation in this study. Patients will be screened and selected from the population of people with strokes who are seen in the Stanford Neuroscience Clinic. Patients will be allowed to participate in any scheduled outpatient rehabilitation during the study. The doctor and/or research coordinator may introduce the study to potential candidates in-person in the Stanford Neurology Clinic, and the research coordinator may contact potential candidates by phone after the doctor's referral.

Procedures:

Once the participant has given informed consent and enrolled in the study, they will have a total of five visits, with one visit every two weeks.

Visit one will entail the participant and identified caregiver undergoing training on the use of the Smart Glove by the research coordinator and Neofect staff. This involves donning/doffing of the glove as well as instruction as to how to use the software program. The participant will be issued a Smart Glove and a tablet preloaded with the software. Subjects will also undergo baseline functional testing, including manual muscle testing (MMT), Fugl-Meyer assessment (FM), Jebsen-Taylor hand function test (JTT), and Stroke Impact Scale (SIS). This first visit is expected to take 60-90 minutes. The participant will be expected to use the Smart Glove for 60 min per day for at least 5 days per week.

The subsequent three visits will be at two week intervals and will involve the participant bringing the device to the Clinical and Translational Research Unit (CTRU). The research coordinator will upload the data from the device as well as troubleshoot any device-related issues. These visits will last 15-30 minutes each.

The final visit will occur after eight weeks of Smart Glove use. In addition to downloading the data, the research coordinator will also repeat functional testing functional testing, including manual muscle testing (MMT), Fugl-Meyer assessment (FM), Jebsen-Taylor hand function test (JTT), and Stroke Impact Scale (SIS). This visit will last 45-60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age 18 and older 2) Diagnosis of stroke at least three months prior to enrollment 3) Unilateral upper extremity functional deficit after stroke 4) Presence of a score of at least 2 points on the medical research council scale for wrist flexion/extension or forearm pronation/supination 5) Able to provide informed consent 6) Caregiver who is willing to be trained in use of the Smart Glove

Exclusion Criteria:

* 1) Predisposing psychological disorders which could impede participation 2) Severe aphasia resulting in communication difficulties 3) Severe pain impeding upper extremity rehabilitation 4) Pre-existing neurological disorder that causes motor deficits (i.e. Parkinson's disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09-23 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2018-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kara Flavin, MD, Principal Investigator — Stanford University; Maarten Lansberg, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital and Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lansberg MG, Legault C, MacLellan A, Parikh A, Muccini J, Mlynash M, Kemp S, Buckwalter MS, Flavin K. Home-based virtual reality therapy for hand recovery after stroke. PM R. 2022 Mar;14(3):320-328. doi: 10.1002/pmrj.12598. Epub 2021 May 24. PMID 33773059

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm - Intervention Arm: RAPAEL Smart Glove Arm used for 8 weeks (60 min per day for at least 5 days per week)
Period: Overall Study
Arm/Group | Single Arm - Intervention Arm
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm - Intervention Arm
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — One patient reported 2 races (Asian and White).
  Participants
    American Indian or Alaska Native | 0
    Asian | 9
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 1
    White | 9
    More than one race | 1
    Unknown or Not Reported | 0
Jebsen Hand Function Test [Mean (Standard Deviation); unit: seconds] — Time (in seconds) to complete the Jebsen-Taylor Hand Function Test. The test consists of 7 subtests. Each subtest is allotted a maximum time of 90 seconds. The Overall Score is the sum of the scores of all seven subtests (max 630 sec). The Fine-Motor Score is the sum of the scores on the four subtests that measure fine-motor function (max 360 sec). The Gross-Motor Score is the sum of the scores on the three subtests that measure gross-motor function (270 sec). Longer time to complete the test indicates worse hand function.
  seconds
    Overall Score | 379 (203)
    Fine-Motor Score | 239 (104)
    Gross-Motor Score | 141 (104)
Fugl-Meyer Assessment [Mean (Standard Deviation); unit: score on a scale] — Score ranges from 0 to 66, with higher scores corresponding to better arm function.
  score on a scale | 41 (11)
Manual Muscle Testing (MMT) Score [Mean (Standard Deviation); unit: score on a scale] — The MMT score is the sum of the Medical Research Council (MRC) scores across 5 domains (elbow flexor, elbow extensor, wrist extension, finger extension and finger flexion) at 8 weeks. Each domain has a scale range of 0 to 5, with higher scores corresponding to better strength. Maximum MMT score ranges from 0-25, with higher scores corresponding to better strength.
  score on a scale | 9.6 (3.3)
Stroke Impact Scale (SIS) [Mean (Standard Deviation); unit: score on a scale] — The score ranges from 0 to 100, with higher scores corresponding to better recovery from stroke.
  score on a scale | 65 (12)

OUTCOME MEASURES:

1. Primary Outcome: Device Use
Description: Number of days during 8 week study-period that patient used the device.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Single Arm - Intervention Arm
Number analyzed (Participants) | 20
days | 27 (34)

2. Secondary Outcome: Device Use Daily Average Per Use Day
Description: Daily average number of minutes of device-use per days that device was used.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Single Arm - Intervention Arm
Number analyzed (Participants) | 20
minutes | 27 (16)

3. Secondary Outcome: Device Use Daily Average
Description: Daily average number of minutes of device-use during 8-week intervention period.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Single Arm - Intervention Arm
Number analyzed (Participants) | 20
minutes | 16.0 (15.4)

4. Secondary Outcome: Jebsen-Taylor Hand Function Test - Overall Score
Description: Time (in seconds) to complete the total Jebsen-Taylor Hand Function Test administered at 8-weeks. The test consists of 7 subtests. Each subtest is allotted a maximum time of 90 seconds. The total score is the sum of the scores of the seven subtests. The total score has a maximum of 630 seconds and there is no minimum. Longer time to complete the test indicates worse hand function.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Single Arm - Intervention Arm
Number analyzed (Participants) | 20
seconds | 353 (208)
Statistical Analysis 1: Comparison: Single Arm - Intervention Arm; Test type: Other; p = 0.025, paired t-test

5. Secondary Outcome: Jebsen-Taylor Hand Function Test - Fine Score
Description: Time (in seconds) to complete the four fine-motor subtests of the Jebsen-Taylor Hand Function Test administered at 8-weeks. Each of the four subtests is allotted a maximum time of 90 seconds. The total score is the sum of the scores of the four subtests. The total score has a maximum of 360 seconds and there is no minimum. Longer time to complete the test indicates worse hand function.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Single Arm - Intervention Arm
Number analyzed (Participants) | 20
seconds | 217 (105)
Statistical Analysis 1: Comparison: Single Arm - Intervention Arm; Test type: Other; p = 0.01, paired t-test

6. Secondary Outcome: Jebsen-Taylor Hand Function Test - Gross Score
Description: Time (in seconds) to complete the three gross-motor subtests of the Jebsen-Taylor Hand Function Test administered at 8-weeks. Each of the three gross-motor subtests is allotted a maximum time of 90 seconds. The total gross-motor score is the sum of the scores of the three subtests. The total score has a maximum of 270 seconds and there is no minimum. Longer time to complete the test indicates worse hand function.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Single Arm - Intervention Arm
Number analyzed (Participants) | 20
seconds | 135 (108)
Statistical Analysis 1: Comparison: Single Arm - Intervention Arm; Test type: Other; p = 0.3, paired t-test

7. Secondary Outcome: Fugl-Meyer Assessment
Description: Upper Extremity Fugl-Meyer Test score at 8-weeks. Score ranges from 0 to 66, with higher scores corresponding to better arm function.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm - Intervention Arm
Number analyzed (Participants) | 20
score on a scale | 43 (12)
Statistical Analysis 1: Comparison: Single Arm - Intervention Arm; Test type: Other; p = 0.098, paired t-test

8. Secondary Outcome: Manual Muscle Testing (MMT) Score
Description: The MMT score is the sum of the Medical Research Council (MRC) scores across 5 domains (elbow flexor, elbow extensor, wrist extension, finger extension and finger flexion) at 8 weeks. Each domain has a scale range of 0 to 5, with higher scores corresponding to better strength. Maximum MMT score ranges from 0-25, with higher scores corresponding to better strength.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm - Intervention Arm
Number analyzed (Participants) | 20
score on a scale | 10.0 (3.4)
Statistical Analysis 1: Comparison: Single Arm - Intervention Arm; Test type: Other; p = 0.2, paired t-test

9. Secondary Outcome: Stroke Impact Scale (SIS)
Description: Score on the SIS at 8-weeks. The score ranges from 0 to 100, with higher scores corresponding to better recovery from stroke.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm - Intervention Arm
Number analyzed (Participants) | 20
score on a scale | 71 (11)
Statistical Analysis 1: Comparison: Single Arm - Intervention Arm; Test type: Other; p = 0.07, paired t-test

10. Secondary Outcome: Patient Experience
Description: Patient self-reported satisfaction with device use (5-point Likert Scale, with higher scores indicating greater satisfaction).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm - Intervention Arm
Number analyzed (Participants) | 20
score on a scale | 4.38 (0.50)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Single Arm - Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-09-23): https://cdn.clinicaltrials.gov/large-docs/29/NCT03559829/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/29/NCT03559829/SAP_001.pdf